CLINICAL TRIAL: NCT00961493
Title: Randomized Controlled Trial of an Acceptance-based Behavior Therapy for Generalized Anxiety Disorder
Brief Title: RCT of an Acceptance-based Behavior Therapy for GAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lizabeth Roemer, Professor of Psychology, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH074589 (NIH); R01MH074589 (NIH); NIH MH074589; DSIR 83-ATAS2
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Acceptance based behavioral therapy
- 2 (Active Comparator)
  Interventions: Behavioral: Applied relaxation

INTERVENTIONS:
Behavioral: Acceptance based behavioral therapy — 16 individual psychotherapy sessions focused on psychoeducation about anxiety, anxious responding, the function of emotions, mindfulness, and problems with efforts to constrict one's emotional experience; training in mindfulness skills; practice applying mindfulness skills in daily life, including acceptance of, rather than efforts to control, internal experience; and identification of values in areas of life and practice engaging in chosen actions.
  Arms: 1
Behavioral: Applied relaxation — 16 sessions of individual psychotherapy focused on psychoeducation about anxiety and anxious responding; training in multiple forms of relaxation; early cue detection; and practice applying relaxation in daily life.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether acceptance-based behavior therapy for GAD results in greater symptom reduction and increased quality of life than applied relaxation.

ELIGIBILITY:
Inclusion Criteria:

* principal diagnosis of GAD
* at least moderate (4 on a scale from 0 to 8) on the ADIS Severity Scale for GAD symptoms
* willing to maintain current psychotropic medication levels (and have been stabilized on any current medications for at least three months) and refrain from other psychosocial treatments for anxiety or mood problems during the course of therapy
* fluent in English
* 18 years or older

Exclusion Criteria:

* bipolar disorder
* psychotic disorders
* substance dependence
* active suicidal intent
* if anxious symptomatology is due to a medical/physical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV, Clinician Severity Rating of GAD | pre-treatment, post-treatment, and 6-, 12-, and 24-month follow-up
Hamilton Anxiety Rating Scale | pre-treatment, post-treatment, and 6-, 12-, and 24-month follow-up
Penn State Worry Questionnaire | pre-treatment, post-treatment, and 6-, 12-, and 24-month follow-up

SECONDARY OUTCOMES:
Beck Depression Inventory - II | pre-treatment, post-treatment, and 6-, 12-, and 24-month follow-up
Quality of Life Inventory | pre-treatment, post-treatment, and 6-, 12-, and 24-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lizabeth Roemer, Ph.D., Principal Investigator — University of Massachusetts, Boston
Locations (1):
- Center for Anxiety and Related Disorders at Boston University, Boston, Massachusetts, United States